CLINICAL TRIAL: NCT06215859
Title: Multi-Center, Randomized, Double-Blind, Placebo (Double-Dummy) and Active-Controlled, Parallel-Group Study of MR-107A-02 for the Treatment of Acute Postoperative Pain Following Herniorrhaphy
Brief Title: Study of MR-107A-02 for the Treatment of Acute Postoperative Pain Following Herniorrhaphy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Specialty LLC (Industry)
Collaborators: Mylan Specialty, LP (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR-107A-02-TFZ-3002
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Pain; Post Operative Pain; Pain
Keywords: Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Pain | interventions — Tramadol; Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MR-107A-02 (Experimental): 15 mg Twice daily (BID) during in patient phase (0-48 hours following randomization) 15 mg BID dosing morning and evening, during out patient phase (5 days) .
  Interventions: Drug: MR-107A-02; Procedure: Herniorrhaphy
- Tramadol (Active Comparator): 50 mg, administered every 6 hours (q6h) during the in patient phase (0-48 hours following randomization).
  Placebo will be administered during out patient phase.
  Interventions: Drug: Tramadol; Drug: Placebo; Procedure: Herniorrhaphy
- Placebo (Placebo Comparator): Placebo is administered every 6 hours (q6h) during the in patient phase (0-48 hours following randomization) and twice daily during the out patient phase.
  Interventions: Drug: Placebo; Procedure: Herniorrhaphy

INTERVENTIONS:
Drug: MR-107A-02 — tablet
  Arms: MR-107A-02
Drug: Tramadol — over-encapsulated tablet
  Arms: Tramadol
Drug: Placebo — over-encapsulated tablet and/or tablet
  Arms: Placebo; Tramadol
Procedure: Herniorrhaphy — Unilateral open inguinal herniorrhaphy with mesh under general anesthesia

SUMMARY:
MR-107A-02 is being studied to investigate its efficacy and safety for treatment of acute pain after herniorrhaphy.

ELIGIBILITY:
Main Inclusion Criteria:

1. Requirement for unilateral open inguinal herniorrhaphy with mesh under general anesthesia.

3. Has an American Society of Anesthesiologists Physical Status of I, II, or III.

4. Pain Intensity (PI) using NRS-R ≥4 at any given timepoint during the 5 hours following end of surgery in the eligibility assessment as well as in the baseline assessment (NRS-R and NRS-A) immediately pre-dosing.

5. Rating of moderate or severe pain on a 4-point categorical pain rating scale (i.e., none, mild, moderate, severe) during the 5 hours following end of surgery.

6. Able to understand and complete the study requirements (including literacy, to enable diary and questionnaire completion), provide written informed consent, and agree to abide by the study protocol and its restrictions.

Main Exclusion Criteria:

1. Previously dosed with this formulation of MR 107A 02.
2. Had any prior inguinal hernia repair in the past 24 months.
3. Has a planned concurrent surgical procedure (e.g., bilateral herniorrhaphy).
4. Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain that is not strictly related to the herniorrhaphy, and which may confound the postoperative assessments.
5. Known hypersensitivity to aspirin, NSAIDs, or other medication used in the study.
6. Body mass index (BMI) >40 kg/m2 at screening.
7. Body weight of <43 kg (105.8 lbs) at screening.
8. History of GI bleeding or peptic ulcer disease.
9. Known active inflammatory bowel disease, e.g., Crohn's Disease or ulcerative colitis.
10. A history of bleeding disorders that may affect coagulation.
11. Subjects with prior stroke or transient ischemic attack in the past 12 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (SPID) for MR-107A-02 versus placebo. | 48 hours after randomization
  SPID based on a 0 to 10-point numeric rating scale with activity (NRS-A) for MR-107A-02 versus placebo.

SECONDARY OUTCOMES:
Number of doses of opioid rescue medication taken for MR-107A-02 versus placebo. | 7 days after randomization
  Number of doses of opioid rescue medication over the combined in-patient and outpatient treatment phases MR-107A-02 versus placebo.
Proportion of subjects using no opioid rescue medication MR-107A-02 versus placebo. | 7 days after randomization
  Proportion of subjects using no opioid rescue medication over the combined in-patient and outpatient treatment phases MR-107A-02 versus placebo.
Summed Pain Intensity Difference (SPID) for tramadol versus placebo. | 7 days after randomization
  SPID based on a 0 to 10-point numeric rating scale with activity (NRS-A) for tramadol versus placebo.
Summed Pain Intensity Difference (SPID) for MR-107A-02 versus tramadol | 48 hours after randomization
  SPID based on a 0 to 10-point numeric rating scale with activity (NRS-A) for MR-107A-02 versus tramadol.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vogt, Study Director — Viatris Inc.
Locations (18):
- United States (18):
  - Investigator site 210, Sheffield, Alabama
  - Investigator site 213, Phoenix, Arizona
  - Investigator site 202, Anaheim, California
  - Investigator site 222, Bakersfield, California
  - Investigator site 208, Riverside, California
  - Investigator site 211, Miami, Florida
  - Investigator site 206, Tampa, Florida
  - Investigator site 207, Atlanta, Georgia
  - Investigator site 205, Wichita, Kansas
  - Investigator site 212, Bellaire, Texas
  - Investigator site 215, Carrollton, Texas
  - Investigator site 204, Houston, Texas
  - Investigator site 216, McAllen, Texas
  - Investigator site 219, San Antonio, Texas
  - Investigator site 203, San Antonio, Texas
  - Investigator site 214, San Antonio, Texas
  - Investigator site 201, Salt Lake City, Utah
  - Investigator site 224, Eau Claire, Wisconsin